CLINICAL TRIAL: NCT05193864
Title: Office-based Validation of the JVPHome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eastern Regional Health Authority (Other)
Collaborators: JVPLabs (Unknown)
Responsible Party: Sponsor
Other Study IDs: 335576
Record Dates: First submitted 2021-11-29; First posted 2022-01-18 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Congestive Heart Failure
Keywords: Remote Monitoring, Machine Vision
MeSH Terms: conditions — Heart Failure | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ambulatory CHF patients: Patients visiting an outpatient CHF clinic
  Interventions: Device: Device: JVPHome and ultrasound

INTERVENTIONS:
Device: Device: JVPHome and ultrasound — Remote clinician assessment of JVP height using the JVPHome, and ultrasound based assessment of JVP height in the same patients.

SUMMARY:
The JVPHome is a novel medical device that utilizes machine vision in order to facilitate assessment of jugular venous pressure (JVP) height relative to the sternal angle with the ultimate goal of enabling remote JVP monitoring. The current study aims to evaluate the ability of an enhanced version of the JVPHome to enable remote identification of JVP height relative to ultrasound among congestive heart failure (CHF) patients when the device is applied by the study team in the clinic.

DETAILED DESCRIPTION:
CHF is a common and devastating health problem estimated to affect upwards of 26 million individuals worldwide. Following an initial hospitalization for heart failure, approximately 25% of patients are readmitted within the first 30 days of discharge. Repeat heart failure hospitalizations are a major burden on both patients and healthcare systems. To date, there is an absence of non-invasive solutions proven to reduce the risk of re-hospitalization for CHF.

The key feature of the physical examination for assessing the volume status of CHF patients is the JVP, which manifests as a biphasic pulsation along the neck. The height of the JVP relative to the sternal angle is a reflection of right atrial pressure, which increases in response to higher pressures transmitted from the left side of the heart. Pathologic elevation of left sided heart pressures can result in fluid congestion in the lungs, which can cause patients to develop shortness of breath and reduced blood oxygen levels. Although a crucial marker of volume status, accurate identification of the JVP can be challenging for physicians due to its pulsations often being subtle.

The JVPHome is a novel medical device designed to facilitate visualization of JVP height relative to the sternal angle through the use of machine vision. The current study aims to evaluate an enhanced version of the JVPHome in a clinic setting when the device is applied to CHF patients by clinicians. Following its application, the JVPHome will be allowed to record a video of the JVP and images will subsequently be transmitted to a secure cloud and undergo analysis with machine vision software. Visualization of the JVP will be facilitated through simultaneous electrocardiographic and pulse oximetry recordings by the JVPHome. Following its application, data is transferred to a secure cloud server for subsequent processing and clinical review.

JVP height of study participants will be concurrently assessed through the use of ultrasound (gold standard). Clinicians that are blinded to ultrasound determined JVP height values will assess JVP height generated by the JVPHome. Analyses will then assess the accuracy of the JVPHome relative to ultrasound and expert clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Congestive heart failure diagnosis receiving ongoing treatment
* Able to provide informed consent

Exclusion Criteria:

* Conditions which preclude visualization of the JVP, including neck deformity, scarring, and facial hair

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Ambulatory CHF outpatients followed at the specialty heart failure clinic at Eastern Health in St. John's, Newfoundland and Labrador, Canada
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-11-03 (Estimated); Study Completion 2023-01-03 (Estimated)

PRIMARY OUTCOMES:
Accuracy of JVP assessment using the JVPHome | Day 1
  Correlation between JVP height assessed by JVPHome and ultrasound Correlation between JVP height assessed by JVPHome and ultrasound Correlation between JVP height assessed by JVPHome and ultrasound

SECONDARY OUTCOMES:
Electrocardiographic Assessment | Day 1
  Evaluate the ability of an embedded ECG sensor to generate a quality single-lead ECG sufficient to identify heart rhythm.
Pulse Oximetry Assessment | Day 1
  Evaluate the ability of an embedded PPG sensor to generate a quality PPG signal in-clinic.
Respiratory Rate | Day 1
  Validate the ability of the JVPHome to measure respiratory rate and compare to expert clinical assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Kris Aubrey-Bassler, MD, Principal Investigator — Eastern Health
Locations (1):
- Eastern Health, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No